

| Study Title | Blended Gaming COVID-19 Training System (BGCTS) with WHO guidelines for staff in residential care homes: A cluster randomised controlled trial |
|---|---|
| Document | BGCTS information sheet |
| Description | |
| Document Date | 11 <sup>th</sup> February, 2021 |
| NCT number | Pending |



## **INFORMATION SHEET**

**Project title:** Blended Gaming COVID-19 Training System (BGCTS) with WHO guidelines for staff in residential care homes: A cluster randomised controlled trial

You are cordially invited to participate in the above project conducted by Dr. Angela Y. M. Leung, School of Nursing, The Hong Kong Polytechnic University. The project has been approved by the Human Subjects Ethics Sub-committee (HSESC) of The Hong Kong Polytechnic University (HSESC Reference Number: HSEARS20200903007).

This study aims to assess the effect of the Blended Gaming COVID-19 Training System (BGCTS) on infection control practices, compliance rates and knowledge of standard precautions among all staff in residential care homes (RCHs).

You will be randomized into either intervention group (IG) or control group (CG). If you are in IG, you will be invited to participate in a 2-week training via a web-based system called BGCTS and attend two face-to-face 30-minute interactive sessions with Infection Control Officer. If you are in CG, you will receive infection control training given by the Infection Control Officer of the RCHs. Before receiving any training in both IG and CG, you will be asked to complete an online quiz and your practice in the RCHs will be observed for two weeks through an on-site camera. After training, you will complete the online quiz and be observed again.

The training should not result in any undue discomfort, but if you feel uncomfortable during the training, you have the right to quit or refuse participation. Observations will be made through the recordings from the cameras which are installed in your workplace. The recordings will be only accessed by the trained research nurse and project team. Your face will be checkered before we conduct the observation, and your name will not be identified in this recording. All faces will be labelled as Staff A, Staff B, etc.

In the online quiz, you will be asked a series of questions about infection control knowledge and practices. No personal identifiers (such as your full name, HK ID number) will be obtained. You will also be assigned a reference number to hide your identity. All information will remain confidential and kept in a secured server/computer/locker and destroyed seven years after the study is completed. Responsible members of The Hong Kong Polytechnic University may be given access for monitoring and/or audit of the research. The Hong Kong Polytechnic University takes reasonable precautions to prevent the loss, misappropriation, unauthorized access or destruction of the information you provide.

If you have any complaints about the conduct of this study, please do not hesitate to contact the Human Subjects Ethics Sub-Committee of The Hong Kong Polytechnic University in writing (c/o Research Office of the University), stating clearly the responsible person and department of this study as well as the HSESC Reference Number.

If you would like more information about this study, please contact XXX via email: XXX

Thank you for your interest in participating in this study.



## CONSENT TO PARTICIPATE IN RESEARCH

| <b>Project Title</b> : Blended Gaming COVID-19 Training System (BGCTS) with WHO guidelines for staff in residential care homes: A cluster randomised controlled trial |
|---|
| hereby consent to participate in the captioned research conducted by XXX. |
| I understand that information obtained from this research will be published. However, my right to privacy will be retained, i.e. my personal details will not be revealed. |
| The procedure as set out in the attached information sheet has been fully explained. I understand the benefit and risks involved. My participation in the project is voluntary. |
| I acknowledge that I have the right to question any part of the procedure and can withdraw at any time without penalty of any kind. |
| Name of participant |
| Signature of participant |
| Name of researcher |
| Signature of researcher |
| Date |